CLINICAL TRIAL: NCT00964210
Title: Prospective Non Controlled Study of Immunogenicity of Human Papilloma Virus (HPV) Vaccine in Groups at Special Risk of Poor Vaccine Result
Brief Title: Protecting Young Special Risk Females From Cervical Cancer Through Human Papilloma Virus (HPV) Vaccination
Acronym: HPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Brockhoff Foundation Australia (Unknown); Shepherd Foundation Australia (Unknown)
Responsible Party: Doctor Jim Buttery, Royal Childrens hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCH CA27091
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2009-08

CONDITIONS: Cervical Cancer
Keywords: Juvenile Idiopathic Arthritis; Inflammatory Bowel Disease; Acute Lymphoblastic Leukemia; Chronic Renal Disease; Solid Organ Transplant
MeSH Terms: conditions — Uterine Cervical Neoplasms; Arthritis, Juvenile; Inflammatory Bowel Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Renal Insufficiency, Chronic | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Licensed quadrivalent HPV vaccine, Gardasil — The dose of the four valent (4v) HPV vaccine is 0.5ml administered by intramuscular (IM)injection. The recommended schedule is 0, 2 and 6 months.

SUMMARY:
A research project is currently being undertaken looking at Human Papilloma Virus (HPV) vaccination in special risk groups. It aims to see if young women with a chronic illness respond well to the HPV vaccine or whether they may require additional doses to ensure protective immunity. The four valent HPV vaccine protects against HPV types 16 & 18, cervical cancer and HPV types 6 & 11, anogenital warts.

The six special risk groups include:

Paediatric Rheumatological Disease Inflammatory Bowel Disease Acute Lymphoblastic Leukaemia Solid Organ Transplant Recipients (kidney and liver) Chronic Renal Disease Bone Marrow Transplants This immunity is measured by antibody levels of the HPV types, which requires a single blood test one month after the final dose of HPV vaccine.

This is compared to healthy controls using antibody response to HPV vaccine. This will assess directly whether these special risk groups respond as well to the HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 12-26 years
* Have been diagnosed by a specialist with one of the six chronic medical conditions described:

  1. Paediatric Rheumatological Disease
  2. Inflammatory Bowel Disease
  3. Acute Lymphoblastic Leukaemia
  4. Solid Organ Transplant Recipients (kidney and liver)
  5. Chronic Renal Disease
  6. Bone Marrow Transplant

Exclusion Criteria:

* Previous immunisation with HPV vaccine Recognised contraindication to the receipt of the vaccine e.g. anaphylaxis

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Determine the HPV vaccine immunogenicity in females 12-26 years with six special risk groups at one month post the third and final HPV vaccination. Blood analysis taken at one month post third and final HPV vaccine to assess immunogenicity. | One Month post HPV vaccination

SECONDARY OUTCOMES:
Describe the safety of the HPV vaccine in the six study groups using self reports and liaison with treating sub specialist team. | One month post third HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jim Buttery, Principal Investigator — NHMRC CCRE in Childhood and Adolescent Immunisation
Locations (1):
- Royal Childrens Hospital, Melbourne, Victoria, Australia